CLINICAL TRIAL: NCT04096001
Title: RCT of Woebot for Substance Use Disorders Phase 1
Brief Title: Woebot for Substance Use Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Woebot Health (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R44DA048712-01 (NIH)
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Results first posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Woebot-SUDs (W-SUDs) — Woebot-SUDs (W-SUDS), an artificially intelligence-powered conversational agent on a smartphone app, eliminates most current SUDs treatment barriers while simultaneously leveraging technology to enhance user experience and engagement. W-SUDs expands and refines existing SUDs treatments by adapting skills from cognitive behavioral therapy, motivational interviewing, and dialectical behavior therapy.

SUMMARY:
Phase 1 of this study aims to develop a digitally-delivered substance use disorder program through the Woebot app-based platform (W-SUDs) and evaluate the effectiveness of, patient satisfaction with and the acceptability of W-SUDs as a substance use management tool.

ELIGIBILITY:
Inclusion Criteria:

* All genders
* 18-65 years
* Must have access to a smartphone and able to download the W-SUDs app
* Committed to engage with app and complete assessments
* Be willing to provide email address (to distribute incentives)
* Be literate in English (as W-SUDs conversational and video materials will be in English)
* Endorse a substance use concern according to the DAST-10 and/or AUDIT-C scale cutoffs for problematic use

Exclusion Criteria:

* Pregnancy (as W-SUDs will not be specifically developed to address the unique needs of this population)
* Suicide attempt or within the past year
* Drug or alcohol overdose within the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Woebot Labs Inc, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Prochaska JJ, Vogel EA, Chieng A, Kendra M, Baiocchi M, Pajarito S, Robinson A. A Therapeutic Relational Agent for Reducing Problematic Substance Use (Woebot): Development and Usability Study. J Med Internet Res. 2021 Mar 23;23(3):e24850. doi: 10.2196/24850. PMID 33755028

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Woebot-SUDs (W-SUDs)
Started | 101
Completed | 51
Not Completed | 50

BASELINE CHARACTERISTICS:
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] — Survey questions: "How old are you?" and "What is your date of birth?"
  years | 36.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Survey question: "What is your biological sex?"
  Participants
    Female | 77
    Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Survey question: "Are you Hispanic or Latinx?"
  Participants
    Hispanic or Latino | 9
    Not Hispanic or Latino | 92
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Survey question following ethnicity question: "Additionally, what best defines your racial background? (select all that apply)
  Participants
    American Indian or Alaska Native | 2
    Asian | 3
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 4
    White | 80
    More than one race | 6
    Unknown or Not Reported | 6
Marital status [Count of Participants; unit: Participants] — Survey question: "Which best describes you?"
  Participants
    Married or cohabitating or partnered | 54
    Divorced or separated or widowed | 14
    Single or never married | 33
Employment status [Count of Participants; unit: Participants] — Survey question: "Which category best describes you?"
  Participants
    Employed full-time | 62
    Employed part-time | 11
    Unemployed, job-seeking | 12
    Other (eg, retired, disabled, homemaker, and student) | 16
COVID-19 situation [Count of Participants; unit: Participants] — Survey question: "What is your current situation with coronavirus/COVID-19? (check all that apply)"
  Participants
    Sheltering in place, lockdown, quarantined | 99
    No restrictions | 2
Lifetime psychiatric diagnoses [Number; unit: participants] — Survey question: "Has a doctor, nurse or other health professional ever told you that you had any of the following mental health conditions? Choose all that apply. If none, please select None."
  participants
    Unipolar depression | 45
    Bipolar or manic depression | 10
    Anxiety disorder | 49
    Posttraumatic stress disorder | 19
    Attention deficit hyperactivity disorder | 15
    Other (eg, obsessive compulsive disorder, eating disorder, and personality disorder) | 12
    Substance use disorder | 6
    Multiple psychiatric diagnoses | 48
    No lifetime psychiatric diagnoses | 28
Therapy experience [Number; unit: participants] — Participants asked about their current therapy situation
  participants
    Never | 30
    Formerly | 45
    Currently | 26
    Currently taking psychiatric medication | 44
Patient Health Questionnaire-8 item depression [Mean (Standard Deviation); unit: units on a scale] — Measure of depression severity. Total score between 0-27, where higher scores indicate greater levels of depression.
  units on a scale | 10.8 (5.8)
General Anxiety Disorder-7 item anxiety [Mean (Standard Deviation); unit: units on a scale] — Measure of anxiety. Total score between 0-21, where higher scores indicate greater levels of anxiety.
  units on a scale | 9.6 (5.7)
Pain intensity in the past 7 days (possible range 0-100) [Mean (Standard Deviation); unit: units on a scale] — Survey questions about current (past 7 days) pain intensity
  units on a scale | 20.4 (22.3)
Pain interfere with normal work in the past 30 days [Count of Participants; unit: Participants] — Survey question about how much a participant's pain has interfered with work during the past 4 weeks
  Participants
    Not at all | 60
    A little bit | 23
    Moderately | 9
    Quite a bit | 7
    Extremely | 2
Primary substance [Count of Participants; unit: Participants] — Participants are provided a list of substances (including alcohol) and asked which substance causes the most problems in their life.
  Participants
    Alcohol | 69
    Cannabis | 20
    Stimulants or cocaine | 7
    Other (eg, club drugs, pain killers, and sedatives) | 5
    Indicated multi-substances | 37
Past 30 days of substance use [Count of Participants; unit: Participants] — Participants provided a list of substances (including alcohol) and asked how many days in the past 30 that they have used each substance
  Participants
    Alcohol | 88
    Cannabis | 50
    Sedatives | 19
    Hallucinogens | 10
    Prescription stimulants | 10
    Cocaine | 5
    Methamphetamine | 4
    Inhalants | 4
    Prescription opioids | 5
    Street opioids | 0
Number of substance use occasions in the past 30 days [Mean (Standard Deviation); unit: occassions] | 31.8 (17.7)
Alcohol Use Disorders Identification Test-Concise [Mean (Standard Deviation); unit: units on a scale] — Survey questions asking participants about their drinking. Population: The overall number of participants analyzed N=101, where n=24 men and n=77 women.
  units on a scale
    Men: number analyzed (Participants) | 24
    Men | 5.2 (3.2)
    Women: number analyzed (Participants) | 77
    Women | 5.5 (3.1)
Drug Abuse Screening Test-10 item [Mean (Standard Deviation); unit: units on a scale] — The DAST-10 is a brief, 10-item self-report assesses consequences related to drug abuse, excluding alcohol and tobacco. The range is 0-10, where higher scores indicate greater severity.
  units on a scale | 3.0 (2.6)
Bothered by cravings in the past 7 days [Count of Participants; unit: Participants]
  Not at all | 7
  A little bit | 31
  Moderately | 33
  Quite a bit | 23
  Extremely | 7
Brief Situational Confidence Questionnaire (BSCQ) [Mean (Standard Deviation); unit: units on a scale] — The 8-item BSCQ is a state dependent measure that assesses self-confidence to resist the urge to drink heavily or use drugs in a variety of situations. Each of the 8 scale situations consists of a 100-mm line, anchored by 0% ("not at all confident") and 100% ("totally confident") where clients are asked to indicate confidence on a scale from 0% to 100%. Higher scores are associated with greater confidence.
  units on a scale | 48.1 (22.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) From Baseline to Post-treatment at 8 Weeks
Description: The AUDIT-C is a widely used 3-item self-report screen for hazardous or harmful alcohol consumption that is based off of the 10-item original AUDIT. The AUDIT-C is scored on a scale of 0-12 (scores of 0 reflect no alcohol use). In men, a score of 4 or more is considered positive; in women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
score on a scale | -9.3 (4.1)

2. Primary Outcome: Change in The Drug Abuse Screening Test 10 (DAST-10) From Baseline to Post-treatment at 8 Weeks
Description: The DAST-10 is a brief, 10-item self-report assesses consequences related to drug abuse, excluding alcohol and tobacco. The range is 0-10, where higher scores indicate greater severity.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
score on a scale | -1.2 (2.0)

3. Primary Outcome: Change in Number of Days Substance Use From Baseline to Post-treatment at 8 Weeks
Description: The number of days a substance was used the past 30 days
Time Frame: Change from Baseline and Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
days | -9.3 (14.1)

4. Secondary Outcome: The Client Satisfaction Questionnaire (CSQ-8) at Post-treatment at 8 Weeks
Description: The CSQ-8 is an 8-item self-report scale measuring satisfaction with treatment. Scores from 8 to 32, with higher values indicating higher satisfaction.
Time Frame: Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
score on a scale | 23.2 (5.5)

5. Secondary Outcome: Usage Rating Profile Intervention (URPI) - Acceptability at Post-treatment at 8 Weeks
Description: URPI-Acceptability Subscale is 6-item subscale from the URP Intervention Revised (URP-IR) scale. The URPI-Acceptability inquires about intervention acceptability. Responses range from 1= "slightly disagree" to 6="strongly agree". Scores are averages, with greater scores indicating greater intervention acceptability.
Time Frame: Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
score on a scale | 25.6 (7.3)

6. Secondary Outcome: Usage Rating Profile Intervention (URPI) - Feasibility at Post-treatment at 8 Weeks
Description: URPI-Feasibility Subscale is 6-item subscale from the URP Intervention Revised (URP-IR) scale. The URPI-Feasibility inquires about factors that impact treatment usage (i.e., intervention quality). Responses range from 1= "slightly disagree" to 6="strongly agree". Scores are averages, with greater scores indicating greater intervention feasibility.
Time Frame: Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
score on a scale | 28.5 (5.7)

7. Secondary Outcome: Change From Working Alliance Inventory (WAI-SR) From Mid-treatment at 4 Weeks to Post-treatment at 8 Weeks
Description: Measure of working alliance. A measure of therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Scores range from 15-60, with higher scores indicating greater alliance. The present study utilized the validated 12-item Short-Revised version (WAI-SR) with minor changes to language, replacing "therapist" with "Woebot".
Time Frame: Change from Mid-treatment at 4 weeks to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
score on a scale | 40.8 (12.5)

8. Secondary Outcome: Change Patient Health Questionnaire (PHQ-8) From Baseline to Post-Treatment at 8 Weeks
Description: Measure of depression severity. Total score between 0-27, where higher scores indicate greater levels of depression.
Time Frame: Change from Baseline to Post-Treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
score on a scale | 8.6 (5.1)

9. Secondary Outcome: Change Generalized Anxiety Disorder (GAD-7) From Baseline to Post-Treatment at 8 Weeks
Description: Measure of anxiety. Total score between 0-21, where higher scores indicate greater levels of anxiety.
Time Frame: Change from Baseline to Post-Treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
score on a scale | -2.3 (4.8)

10. Secondary Outcome: Change Brief Situational Confidence Questionnaire (BSCQ) From Baseline to Post-Treatment at 8 Weeks
Description: The 8-item BSCQ is a state dependent measure that assesses self-confidence to resist the urge to drink heavily or use drugs in a variety of situations. Each of the 8 scale situations consists of a 100-mm line, anchored by 0% ("not at all confident") and 100% ("totally confident") where clients are asked to indicate confidence on a scale from 0% to 100%. Higher scores are associated with greater confidence.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
units on a scale | 16.9 (21.4)

11. Secondary Outcome: Change Pain Rating From Baseline to Post-Treatment at 8 Weeks
Description: Range from 0-100 (no pain to worst pain imaginable).
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Woebot-SUDs (W-SUDs)
Number analyzed (Participants) | 51
score on a scale | 24.2 (22.0)

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed at post-treatment, 8 weeks from baseline.
Description: Serious adverse events occurring during treatment were assessed for hospitalization related to substance use, suicide attempt, alcohol or drug overdose, and severe withdrawal (eg, delirium tremens). Positive endorsements were followed up with questions about the timing, diagnosis, and resolution. If additional details were needed to determine whether the event was study related, a team member reached out to the participant.
Arm/Group | Woebot-SUDs (W-SUDs)
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 1/101
Other Adverse Events (participants affected / at risk) | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Woebot-SUDs (W-SUDs) (N=101)
Sepsis (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT04096001/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT04096001/SAP_002.pdf
  • Informed Consent Form (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT04096001/ICF_000.pdf